CLINICAL TRIAL: NCT00631982
Title: In Vitro Maturation of Oocytes for Patients With Polycystic Ovaries
Brief Title: Invitro Maturation of Oocytes for Patients With Polycystic Ovaries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: IVF and Infertility Unit, Assaf Harofeh Medical Center, Zerifin Israel, Assaf Harofeh Medical Center, Zerifin Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22/08
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-03

CONDITIONS: Infertility; Polycystic Ovaries
Keywords: in vitro maturation oocytes
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome

ARMS (1):
- Group I (Experimental): patients with PCO undergoing in vitro maturation and subsequently IVF and embryo transfer
  Interventions: Procedure: in vitro matuartion of oocytes

INTERVENTIONS:
Procedure: in vitro matuartion of oocytes — in vitro maturation of (immature) oocytes

SUMMARY:
In vitro maturation of oocytes after minimal gonadotropin stimulation in patients with polycystic ovaries, to prevent cases of ovarian hyperstimulation.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovaries
* Needing IVF for fertility treatment

Exclusion Criteria:

* Age above 39

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
maturation rate, | 18 months

SECONDARY OUTCOMES:
Fertilization rate, pregnancy rate | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- IVF and Infertility Unit, Assaf Harofeh Medical Center, Ẕerifin, Israel